CLINICAL TRIAL: NCT07077187
Title: Effect of Rasagiline on Balance in Parkinson's Disease as Measured by Computerized Posturography
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding for the study could not be obtained.
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Robert Fekete, Associate Professor, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-10,768
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: balance; posturography; computerized dynamic posturography; rasagiline; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Intervention Model Description: The study will test the hypothesis that therapy with rasagiline improves balance in PD patients as measured by computerized dynamic posturography. 5 subjects will be randomized to rasagiline or placebo and 5 further subjects will be randomized to rasagiline as adjuvant therapy versus placebo. Subjects will be analyzed by computerized dynamic posturography testing. The device measures body sway under varying visual and vestibular cues and is used for assessment of balance. Subjects will be evaluated at baseline prior to taking first tablet as well as at 4 weeks and 8 weeks. In the adjuvant therapy arm, subjects will be evaluated on rasagiline but in a functional OFF state for their other PD medications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rasagiline monotherapy (Active Comparator): Participants will be taking rasagiline 1 mg oral tablet daily
  Interventions: Diagnostic Test: computerized dynamic posturography; Drug: Rasagiline 1 mg capsule
- placebo monotherapy (Placebo Comparator): Participants will be taking placebo 1 mg orally daily.
  Interventions: Diagnostic Test: computerized dynamic posturography; Drug: Placebo
- rasagiline adjuvant therapy (Active Comparator): Participants will be taking rasagiline 1 mg orally daily as adjuvant therapy in addition to their stable existing Parkinson disease medication.
  Interventions: Diagnostic Test: computerized dynamic posturography; Drug: Rasagiline 1 mg capsule
- placebo adjuvant therapy (Placebo Comparator): Participants will be taking placebo 1 mg orally daily as adjuvant therapy in addition to their stable existing Parkinson disease medication.
  Interventions: Diagnostic Test: computerized dynamic posturography; Drug: Placebo

INTERVENTIONS:
Diagnostic Test: computerized dynamic posturography — Patients in each arm will have computerized dynamic posturography performed at baseline prior to taking first tablet as well as at 4 weeks and 8 weeks. In the adjuvant therapy arm, subjects will be evaluated on rasagiline but in a functional OFF state for their other Parkinson disease medications.
Drug: Rasagiline 1 mg capsule — Rasagiline 1 mg oral tablet daily will be administered to study participants.
  Arms: Rasagiline monotherapy; rasagiline adjuvant therapy
Drug: Placebo — Placebo 1 mg oral tablet daily will be administered to study participants.
  Arms: placebo adjuvant therapy; placebo monotherapy

SUMMARY:
This study evaluates the effect of rasagiline on balance in Parkinson's disease. Participants taking study medication which is rasagiline or sugar pill will undergo a computerized balance test on and off medication. Participants will stand on a platform which which moves slightly and a computer will measure their body sway and provide a balance score.

DETAILED DESCRIPTION:
The study will test the hypothesis that therapy with rasagiline improves balance in PD patients as measured by computerized dynamic posturography. 5 subjects will be randomized to rasagiline or placebo and 5 further subjects will be randomized to rasagiline as adjuvant therapy versus placebo. Subjects will be analyzed by computerized dynamic posturography testing. The device measures body sway under varying visual and vestibular cues and is used for assessment of balance

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or above
2. Clinical diagnosis of Parkinson disease by verified by movement disorders expert at the initial study visit with at least two cardinal signs of the disease (rest tremor, bradykinesia, rigidity, and postural instability).
3. For the monotherapy arm, patients must not be on amantadine, dopamine agonists, or levodopa. For the adjuvant therapy arm: Patients must be on a stable dose of their current medication for treatment of Parkinson disease which may include any combination of the following: amantadine, trihexiphenydil, dopamine agonist, and/or levodopa.
4. Patients may continue their stable dose of tricyclic, selective serotonin reuptake inhibitor, or serotonin norepinephrine reuptake inhibitor if they are on these medications at randomization.

Exclusion Criteria:

1. Catechol-O-Methyltransferase (COMT) inhibitor therapy use 30 days prior to start of study (both study arms).
2. Dopamine receptor blocker use (such as quetiapine) one week prior to taking study drug
3. For both monotherapy and adjuvant therapy arms: use of MAO inhibitor therapy including selegiline or rasagiline within 30 days prior to taking study drug and first posturography evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Computerized Dynamic Posturography Strategy Composite Score | 8 weeks
  Change from baseline to week 8 measurement of Computerized Dynamic Posturography Strategy Composite Score will be compared among the 4 arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fekete, MD, Principal Investigator — New York Medical College

IPD SHARING:
Plan to Share IPD: No
Institutional Review Board approval explicitly marked clinical study data as protected patient data and stated that data will be stored locally.

REFERENCES:
- [Background] Ondo WG, Almaguer M, Cohen H. Computerized posturography balance assessment of patients with bilateral ventralis intermedius nuclei deep brain stimulation. Mov Disord. 2006 Dec;21(12):2243-7. doi: 10.1002/mds.21165. PMID 17078067

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-09-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT07077187/Prot_SAP_ICF_001.pdf